CLINICAL TRIAL: NCT02308423
Title: Clinical and Radiologic Follow up of Subchondral Fractures of the Glenoid
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0204-14-MMC
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Subchondral Fractures of the Glenoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: XR of shoulder — Radiologic examination: Axial view, Axillary view and Anterior posterior view- to evaluate the level of osteoarthritis by Kellgren Lawrence score and Samilson score.

SUMMARY:
in this study the investigators will call patients who had Subchondral fractures and treated in our department over the last 20 years.

The investigators will evaluate their shoulder function by a questionary, Constant score and radiologic evaluation.

DETAILED DESCRIPTION:
Patient evaluation by:

- Physical examination, questionary Constant score: Pain (severe, moderate, mild, non), activity level (sleep affected/sport limitations/daily living limitations/arm positioning) and range of motion (forward flexion/lateral elevation, internal and external rotation).

- Radiologic examination: Axial view, Axillary view and Anterior posterior view- to evaluate the level of osteoarthritis by Kellgren Lawrence score and Samilson score.

ELIGIBILITY:
Inclusion Criteria:

* Any man or women who had subchondral fractures of the glenoid

Exclusion Criteria:

* Pregnant women
* Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients 18-80 yo who had subchondral fractures of the glenoid
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Function disability of the shoulder | 20 years
  The patients will be invited to the clinic where the investigators will examine them and define a "constant score" that takes in consideration: Pain, Activity level and Range of motion.

SECONDARY OUTCOMES:
Measurement of degenerative changes of the gleno-humeral joint. | 20 years
  The investigators will assess the status of osteoarthrosis of the gleno-humeral joint, this will be measured by the Kellgren Lawrence (0-4) and the Samilson (0-3) scores.